CLINICAL TRIAL: NCT07284186
Title: A Phase 1, First-in-Human Study of the SMARCA2 Degrader, PLX-61639, in Patients With SMARCA4-Mutated Locally Advanced or Metastatic Solid Tumors
Brief Title: First-in-Human Study of PLX-61639 in Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Plexium, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PLX-61639-101
Record Dates: First submitted 2025-11-20; First posted 2025-12-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Squamous Cell Carcinoma; Gastric Adenocarcinoma; Gastric Squamous Cell Carcinoma; Gastroesophageal Junction (GEJ) Adenocarcinoma; Metastatic Solid Tumor; Non-Small Cell Lung Carcinoma; Esophageal Adenocarcinoma; SMARCA4 Mutation; Gastroesophageal Junction Squamous Cell Carcinoma; Advanced Solid Tumor
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Adenocarcinoma; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Intervention Model Description: In Part 1, eligible participants will enroll sequentially in up to 5 escalating PLX-61639 dose cohorts.
  In Part 2, participants will be randomized 1:1 to 1 of 2 dose levels at or below the maximally tolerated (or administered) dose evaluated during Part 1.
  In Part 3, additional participants will enroll sequentially to 1 dose level selected from Part 2.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PLX-61639 (Experimental)
  Interventions: Drug: PLX-61639

INTERVENTIONS:
Drug: PLX-61639 — Orally available degrader of SMARCA2

SUMMARY:
A multicenter, single-arm, first-in-human study to investigate the safety, pharmacokinetics, and preliminary antitumor activity of PLX-61639 in participants with locally advanced or metastatic, relapsed/refractory, SMARCA4-deficient solid tumors who are intolerant of or have failed available, approved therapies.

The study will be conducted in 3 parts: dose escalation (Part 1), dose optimization (Part 2), and cohort expansion (Part 3). Each part of the study will consist of a Screening Phase lasting up to 28 days during which participants will be assessed for eligibility, a Treatment Phase beginning on Cycle 1 Day 1 and consisting of consecutive 28-day cycles, an End of Treatment Visit, and a Post-Treatment Follow-Up Phase.

Participants will receive their assigned dose of PLX-61639 administered orally, once daily until progression/relapse, intolerance, death, or withdrawal from study treatment by the Investigator or participant.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with locally advanced or metastatic, relapsed/refractory, solid tumors harboring a SMARCA4 loss-of-function mutation that have progressed on, are intolerant of, or not otherwise candidates for available approved therapies
* Adequate liver bone marrow, coagulation, renal, and cardiopulmonary function
* Measurable disease per RECIST 1.1
* ECOG PS of 0 or 1

Key Exclusion Criteria:

* Germline SMARCA4 mutations
* Known SMARCA2 mutation or loss of expression
* Symptomatic CNS disease
* Prior treatment with another SMARCA2-directed therapy
* History of other malignancies
* Clinically significant heart disease
* Uncontrolled hypertension
* Prolongation of QT interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events | From enrollment to 28 days after the last dose of PLX-61639
Dose-Limiting Toxicities | From enrollment to 28 days after first dose of PLX-61639

SECONDARY OUTCOMES:
Dose reductions due to Adverse Events | From Day 1 to the end of PLX-61639 treatment, an average of 1 year
Study treatment discontinuations for reasons other than disease progression | From Day 1 to the end of PLX-61639 treatment, an average of 1 year
Pharmacokinetics of PLX-61639: Cmax | From Day 1 to Day 15 of Cycle 1 (Part 1 only) (each cycle is 28 days)
Pharmacokinetics of PLX-61639: Tmax | From Day 1 to Day 15 of Cycle 1 (Part 1 only) (each cycle is 28 days)
Pharmacokinetics of PLX-61639: AUC0-last | From Day 1 to Day 16 of Cycle 1 (Part 1 only) (each cycle is 28 days)
Radiographic response to PLX-61639 | From Day 1 to the end of PLX-61639 treatment, an average of 1 year
Time to response (TTR) to PLX-61639 | From Day 1 to achievement of partial or complete response, up to 24 weeks
Duration of response (DoR) to PLX-61639 | From first documented partial or complete response to disease progression or death, an average of 1 year
Progression Free Survival (PFS) of PLX-61639 | From Day 1 to disease progression or death, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Plexium, Inc.
Locations (10):
- United States (10):
  - Research Site, Scottsdale, Arizona
  - Research Site, Duarte, California
  - Research Site, Orange, California
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, San Antonio, Texas
  - Research Site, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No